CLINICAL TRIAL: NCT05681845
Title: A Study to Demonstrate Bioequivalence of a Single Subcutaneous Administration of NNC0365-3769 (Mim8) With the DV3407-C1 Pen Injector Versus a Syringe and Enhanced Cartridge in Healthy Male Participants
Brief Title: A Study to Compare the Blood Levels of Mim8 in Healthy Men When Administered With the DV3407-C1 Pen Injector or a Syringe and Cartridge
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NN7769-4992; U1111-1277-9765 (Other: World Health Organization (WHO)); 2022-002318-18 (EudraCT Number)
Record Dates: First submitted 2023-01-04; First posted 2023-01-12 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Haemophilia A
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The study consists of two parts - an open-label pilot part and a double-blind bioequivalence part.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Arm 1 (Pilot part) (Experimental): Participants will receive a single dose of Mim8 using a 32G, 4 mm pen-needle with the DV3407-C1 pen injector.
  Interventions: Drug: NNC0365-3769 (Mim8)
- Arm 2 (Pilot part) (Experimental): Participants will receive a single dose of Mim8 using a 29G, 8 mm needle and syringe with the enhanced cartridge.
  Interventions: Drug: NNC0365-3769 (Mim8)
- Arm 3 (Bioequivalence part) (Experimental): Participants will receive a single dose of Mim8 using a 29G, 4 mm pen-needle with the DV3407-C1 pen injector.
  Interventions: Drug: NNC0365-3769 (Mim8)
- Arm 4 (Bioequivalence part) (Experimental): Participants will receive a single dose of Mim8 using a 29G, 8 mm needle and syringe with the enhanced cartridge.
  Interventions: Drug: NNC0365-3769 (Mim8)

INTERVENTIONS:
Drug: NNC0365-3769 (Mim8) — Participants will receive a single dose of Mim8 subcutaneously in the abdomen.

SUMMARY:
Novo Nordisk is developing the study medicine Mim8 for the treatment of haemophilia A. The study aims to show similar levels of Mim8 in blood when using a new pen injector, called DV3407-C1 pen injector, and when using a syringe and cartridge. The new pen injector is intended to facilitate the administration of Mim8 for patients with haemophilia A. The participants will get Mim8 as injection under the skin (subcutaneously) of the belly using the DV3407-C1 pen injector and a needle (hereinafter referred to as pen injector) or using a needle and syringe from a cartridge (hereafter called syringe and cartridge). The participants will receive one injection with Mim8, either with the DV3407-C1 pen injector or with a syringe and cartridge. The study participation will last up to 20 weeks. Only healthy men can take part in the study.

ELIGIBILITY:
Inclusion Criteria:

* Male aged 18-55 years (both inclusive) at the time of signing informed consent.
* Body mass index (BMI) between 18.5 and 29.9 kilogram per square metre (kg/m^2) (both inclusive) at screening.
* Body weight between 60.0 and 100.0 kg (both inclusive) at screening.
* Considered to be generally healthy based on the medical history, physical examination, and the results of vital signs, electrocardiogram and clinical laboratory tests performed during the screening visit, as judged by the investigator.

Exclusion Criteria:

* Increased risk of thrombosis, e.g., known history of personal or first-degree relative(s) with unprovoked deep vein thrombosis.
* Any clinical signs or established diagnosis of venous or arterial thromboembolic disease.
* Factor VIII activity greater than or equal to (≥) 150 percent (%) at screening.
* Thrombophilia as identified by any of the below laboratory markers at screening:
* Protein C, protein S or antithrombin less than (<) lower limit of normal (LLN)
* Factor II activity or activated protein C resistance >upper limit of normal (ULN).

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 205 (Actual)
Dates: Start 2023-01-02 (Actual); Primary Completion 2023-10-13 (Actual); Study Completion 2023-10-13 (Actual)

PRIMARY OUTCOMES:
AUC0-112 days, SD: area under the Mim8 plasma concentration-time curve from time 0 until 112 days after a single dose | From time of dosing (day 1) to day 113
  Measured in micrograms*day per milliliter (μg*day/mL).
Cmax, SD: maximum plasma concentration of Mim8 after a single dose | From time of dosing (day 1) to day 113
  Measured in μg/mL.

SECONDARY OUTCOMES:
AUC0-inf, SD: area under the Mim8 plasma concentration-time curve from time 0 to infinity after a single | From time of dosing (day 1) to day 113
  Measured in μg*day/mL.
t1/2, SD: the terminal half-life of Mim8 after a single dose | From time of dosing (day 1) to day 113
  Measured in days.
tmax, SD: the time to maximum concentration of Mim8 after a single dose | From time of dosing (day 1) to day 113
  Measured in days.
Number of injection site reactions | From time of dosing (day 1) to day 113
  Measured in count of events.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (1):
- Charité - Campus Charité Mitte - Charité Research Organisation GmbH, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com